| Prospective Randomized comparison Of prosthetic Valve Effective |
|------------------------------------------------------------------|
| orifice area: One-year analysis of two bovine PERIcardial valves |
| (PROVE-PERI trial) |

NCT 03796442

Trial Protocol v 1.4

Updated Dec 28, 2018

**Statistical Analysis Plan** 

1. Inclusion criteria

Patients who are scheduled to undergo AVR

② Over 19 years of age

3) Patients who are planned to receive a bioprosthetic valve for aortic valve substitute

4 Patients who or whose legal representative fill out a written consent form before the start

of the clinical trial and patients who can comply with the clinical trial requirements

2. Exclusion criteria

1) Patients with concomitant mitral or tricuspid valve operation

Patients with severe left ventricular dysfunction (ejection fraction < 0.30)

3 Patients with infective endocarditis

4 Patients with a medical history such as a malignant disease that might limit the possibility

of mid-term follow-up

5 Patients who refused study enrollment

3. Sample size calculation

The study is designed to have 80% power to detect 1-year AVMPG of 12.6±4.3mmHg for the

study prosthesis [1] and 11.9±4.3mmHg for the control prosthesis, [2] with a 1-sided type I error

of 2.5% and a noninferiority margin of 3mmHq. The noninferiority margin was determined by

the values of 15mmHg for AVMPG of clinically significant aortic stenosis [3] and 12mmHg for

AVMPG of the control prosthesis. Fifty-six patents in each group were needed to complete the

study cohort. Allowing for a 20% dropout rate during the 1-year follow-up, we determined that

the recruitment of 70 patients in each group was necessary.

(1) Level of significance ( $\alpha$ ) = 0.025

(2) Type II error ( $\beta$ ) = 0.20, power of the test = 80%

(3) Drop out rate = 20%

(4) One-tailed test

 $H_0$ (null hypothesis):  $\mu_1 - \mu_2 \geq \delta$ 

 $H_1$ (alternative hypothesis):  $\mu_1 - \mu_2 < \delta$ 

2

( $\mu_1$ : mean AVMPG of the study group on 1 – year echocardiographic follow – up ,  $\mu_2$ : mean AVMPG of the control group on 1 – year echocardiographic follow – up  $\delta$ : noninferiority margin)

The calculation was performed using PASS Software(Power Analysis and sample size software: http://www.ncss.com), and the calculated formula is as follows.

$$n = \frac{\left(Z_{\alpha} + Z_{\beta}\right)^2 ({\sigma_1}^2 + {\sigma_2}^2)}{\left((\mu_1 - \mu_2) - \delta\right)^2}$$

 $\mu_1 = \text{mean AVMPG}$  of the study group on 1-year echocardiographic follow -up

 $\mu_2 = \text{mean AVMPG}$  of the control group on 1 - year echocardiographic follow - up

 $\sigma_1$  = standard deviation of AVMPG of the study group on 1 – year echocardiographic follow – up

 $\sigma_2$  = standard deviation of AVMPG of the control group on 1 – year echocardiographic follow – up

 $\delta$ : noninferiority margin

- Primary clinical endpoint mean pressure gradient across the aortic valve (AVMPG) on 1-year echocardiographic follow-up
- Secondary clinical endpoint
  the effective orifice area (EOA) on 1-year echocardiographic follow-up
  operative mortality, operative morbidities
  1-year clinical outcomes (all-cause mortality, cardiac death and major adverse events)

The primary endpoint of the PROVE-PERI trial is AVMPG on 1-year echocardiographic follow-up. The secondary endpoints are the EOA on 1-year echocardiographic follow-up and 1-year clinical outcomes including all-cause mortality, cardiac death and MAEs.

The study is designed to have 80% power to detect 1-year AVMPG of 12.6±4.3mmHg for the study prosthesis [2] and 11.9±4.3mmHg for the control prosthesis, [4-6] with a 1-sided type I error of 2.5% and a noninferiority margin of 3mmHg. The noninferiority margin is determined by the values of 15mmHg for AVMPG of clinically significant aortic stenosis [7] and 12mmHg for AVMPG of the control prosthesis. Fifty-six patents in each group are needed to complete the study cohort. Allowing for a 20% dropout rate during the 1-year follow-up, we determine that the recruitment of 70 patients in

each group was necessary.

Statistical analyses will be performed using SPSS software (version 25.0; IBM, Armonk, NY) and SAS software (version 9.3; SAS Institute, Cary, NC). Data will be expressed as the mean ± standard deviation, median with IQRs or proportions. Comparisons between the 2 groups will be made using the chisquare test and Fisher's exact test for categorical variables and Student's t-test or the Mann–Whitney test for continuous variables, as appropriate. The null hypothesis is that the Avalus<sup>TM</sup> is inferior to the CEPME based on the AVMPG at 1-year echocardiographic follow-up, with a non-inferiority margin of 3mmHg. The result for the primary endpoint is presented with 97.5% one-sided confidence interval for mean difference between groups. The non-inferiority test will be performed using a t-test which compares mean difference between groups with the non-inferiority margin under the one-sided significance level of 0.025. For analysis of 1-year clinical outcomes including all-cause mortality, cardiac death, and MAEs, events will be counted at postoperative 1 year, and comparisons between the 2 groups will be made using the chi-square test and Fisher's exact test. A P value of < .050 will be considered statistically significant. All outcomes will be compared with an intention-to-treat base. Perprotocol and as-treated analyses will be added for hemodynamic outcomes.

## References

- 1. Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, et al. 2017 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2017;38:2739-2791.
- 2. Klautz RJM, Kappetein AP, Lange R, Dagenais F, Labrousse L, Bapat V, et al. Safety, effectiveness and haemodynamic performance of a new stented aortic valve bioprosthesis. Eur J Cardiothorac Surg. 2017;52:425-431.
- 3. D Rennie. How to report randomized controlled trials. The CONSORT statement. JAMA. 1996;276:649.
- 4. Fiegl K, Deutsch MA, Rondak IC, Lange R, Guenzinger R. Matched Comparison of Two Different Biological Prostheses for Complete Supra-annular Aortic Valve Replacement. Thorac Cardiovasc Surg.

2015;63:459-66.

- 5. Wendt D, Thielmann M, Plicht B, Aßmann J, Price V, Neuhäuser M, et al. The new St Jude Trifecta versus Carpentier-Edwards Perimount Magna and Magna Ease aortic bioprosthesis: is there a hemodynamic superiority? J Thorac Cardiovasc Surg. 2014;147:1553-60.
- 6. Wyss TR, Bigler M, Stalder M, Englberger L, Aymard T, Kadner A, et al. Absence of prosthesis-patient mismatch with the new generation of Edwards stented aortic bioprosthesis. Interact Cardiovasc Thorac Surg. 2010;10:884-7.
- 7. Baumgartner H, Hung J, Bermejo J, Chambers JB, Evangelista A, Griffin BP, et al. Echocardiographic assessment of valve stenosis: EAE/ASE recommendations for clinical practice. Eur J Echocardiogr. 2009;10:1-25.